CLINICAL TRIAL: NCT03788460
Title: A Retro-prospective Pediatric Data Collection Study of the Correlation Between PT and the Level of Coagulant Factor VII
Brief Title: Correlation Between PT and INR to Factor 7
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Laniado Hospital (Other)
Responsible Party: Principal Investigator, Dr. Nechama Sharon, Head, Pediatric hemato-oncology unit, Laniado Hospital
Other Study IDs: 0062-18-LND
Record Dates: First submitted 2018-12-11; First posted 2018-12-27 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Epistaxis; ENT Disorder
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- childrens population with lack of Factor VI: We will check PT levels, we will concentrate the data in the table, along with personal information such as age and gender.
  We will try to conduct a statistical relationship between the PT values and Factor VII levels, to look for statistical significance, we will try to find a model for predicting the level of factor VII based on PT
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The purpose of our study:

Given the large number of coagulability tests done before a number of surgeries, specially otolaryngology procedures, such as tonsillectomy and adenoidectomy, as well as a part of epistaxis workup, prothrombin time (PT) and partial thromboplastin time (PTT) were checked, and it was found that in some people there is an isolated elongated PT, a low level of factor VII was found in these people.

The purpose of the current study is to find a correlation between the value of PT\INR and the level of factor VII, we tried to do so by a retro-prospective study on patients known to have a factor VII deficiency at Laniado hospital, such a correlation could make both the diagnosis and the management of people with factor VII deficiency easier and more accessible.

The study levels:

1. Data collection : On the children's population who are known for their lack of Factor VII, we will check PT levels, we will concentrate the data in the table, along with personal information such as age and gender
2. Data Processing : We will try to conduct a statistical relationship between the PT values and Factor VII levels, to look for statistical significance, we will try to find a model for predicting the level of factor VII based on PT

Number of participants:

60 participants

Ages of participants:

0-18 years old

Gender of participants:

Both sexes

Inclusion criteria:

1. A participant who is 0-18 years old
2. A participant who is, except for bleeding tendency, healthy in general
3. A participant who has elongated PT
4. A participant who has normal PTT

Exclusion criteria:

1. Background disease
2. Use of medications
3. Use of anti coagulation drugs

The duration of the study :

The study is of a retrospective type, we already have a number of subjects, we need more as to reach statistical significance, so the expectation is two to three months

DETAILED DESCRIPTION:
Factor VII is one of the main components of the coagulation process. It belongs to the serine proteases and it dependents on vitamin K in order to function. Its primary function is to initiate the clotting process itself, along with tissue factor: Following a vascular endothelial injury, there is a response of vasoconstriction, the blood flow in contact with the subendothelial matrix, at that time, TF, a protein in the same matrix, binds to and activates the VII coagulation factor, then, FVIIa-TF complex begins the coagulation cascade, at the end of that cascade, fibrin is formed.

The factor VII gene is located on the long arm of chromosome 13, sized 12 kD, contains 12 axons that encode a protein composed of 406 amino acids, it's located at a distance of 2.8 kD from the gene of factor X.

More than 120 mutations have been found in factor VII gene to date, the association between genotype and phenotypes is unclear in most cases however. Seligsohn and his colleagues described one of the mutations in Factor VII, 5-Ser339Phe, which was found in three Tunisian families and caused a tendency to bleed through a mechanism of reduced factor X activation.

When it comes to Factor VII deficiency, the missing is never hermetic as such condition is not compatible with life as seen from work on knockout mice. Partially missing factor VII is the most common of all rare coagulation problems. Clinically, these are usually epistaxis, easy bruising, gum bleeding, muscle hematoma, hamarhtrosis, hematuria, postoperative bleeding, although there may also be conditions of life threatening blood in the nervous system and in the gastrointestinal tract. Except for increased menstruation that occurs in about 70% of the women with factor VII deficiency, there is no gender difference in symptoms.

Suspicion of Factor VII deficiency is usually done in the course of screening in family members with a known deficiency or on tests following an episode of bleeding, such as epistaxis or surgery in areas with a tendency to bleed (nose, throat or teeth) .

An abnormal PT test indicates a lack of factor VII. An elongated PTT test can suggest hemophilia A and B (missing factors VIII and IX, respectively), lack of factor XI, incomplete factor XII or von disease willebrand / VWF . The extension of PT also implies a deficiency in the factors X, V, II and fibrinogen, and the result is represented by a percentage relative to normal people.

The diagnosis of Factor VII deficiency is laboratory. The initial laboratory tests are PT, aPTT and platelet count, followed by a FVII coagulant activity test for prolonged PT states. In order to confirm the result, the FVII assay is performed again

Prothrombin time is typically analyzed by a laboratory technologist on an automated instrument at 37 °C. Blood is drawn into a test tube containing liquid sodium citrate, which acts as an anticoagulant by binding the calcium in a sample. The blood is mixed, then centrifuged to separate blood cells from plasma (as prothrombin time is most commonly measured using blood plasma). A sample of the plasma is extracted from the test tube and placed into a measuring test tube Next an excess of calcium is added to the test tube, thereby reversing the effects of citrate and enabling the blood to clot again. Finally, in order to activate the extrinsic / tissue factor clotting cascade pathway, tissue factor is added and the time the sample takes to clot is measured optically. The prothrombin ratio (INR) is the prothrombin time for a patient sample divided by the result for control plasma.

There are two types of Factor VII deficiency. The first is a quantitative with both a lack of FVII coagulant activity and with a low level of FVII antigen, the second one is qualitative with a low FVII coagulant activity but a normal level of FVII antigen. In fact, the examination of the antigen distinguishes between these two missing types, but does not predict the tendency to bleed, and it is not recommended to diagnose Factor VII deficiency on the basis of the antigen test. However, for known patients receiving a recombinant factor it can be useful.

There are no clear guidelines for the treatment of hereditary deficiency VII. Recombinant factor VII is a choice in many cases for both children and adults, but there are other treatment options as discussed in our study.

The purpose of the current study is to find a correlation between the value of PT\INR and the level of factor VII, we tried to do so by a retro-prospective study on patients known to have a factor VII deficiency at Laniado hospital, such a correlation could make both the diagnosis and the management of people with factor VII deficiency easier and more accessible.

ELIGIBILITY:
Inclusion Criteria:

Elongated PT value; Normal PTT value;

-

Exclusion Criteria:

Background medical conditions; Taking anticoagulants; Taking chronic medications;

-

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with known factor VII deficiency
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-07 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between PT, INR and the level of coagulant factor VII | Study completion within 2 years
  correlation between PT / INR value and percent of factor VII through a retro-prospective study of patients who are known to have factor VII deficiency. This correlation is expected to facilitate diagnostic and monitoring procedures for patients with factor VII deficiency. The clinical value of this study is to facilitate diagnosis and treatment in patients with Factor VII defiency.

IPD SHARING:
Plan to Share IPD: No